CLINICAL TRIAL: NCT07043309
Title: Study the Diagnostic and Therapeutic Role of Flexible Bronchoscopy in the Patients Attending Assuit University Children Hospita
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Gamal Darwish, residant doctor at Assiut university, Assiut University
Other Study IDs: diagm/therap bronchoscopy
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Chest Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: All children in pediatric bronchoscopy unit

SUMMARY:
Bronchoscopyhasbeenutilizedinchildrenforlongforthediagnosisofairwayabnormalitiesand obtainingbronchoalveolarlavage.Thoughtherehasbeenrapidgrowthofbronchoscopic interventionsinadultpatients,useinchildrenhasbeenlimited.Newerbronchoscopictechnologies andinstrumentsarefocussedlargelyonadultpatients.Riskofsedationandsmallairwaysizealso havebeenlimitingfactors.Butrecentadvancesinequipmentsintheformofhinnerbronchoscopes withworkingchannelsandthinnerinstrumentshavefacilitatedbronchoscopicinterventionsin children.(1) Pediatricflexiblelaryngotrachealbronchoscopy(FB)isahighlyversatileandeffectivediagnostic andtherapeutictoolwithanimportantroleinpediatricrespiratorymedicine. Itwasfirstdescribedin 1968andappliedinthepediatricpopulation10yearslater.(2,3,4) Nowadays,FBisanintegralpartofthemaagementofneonates, infants,andchildrenwithvarious lungandairwaydiseases. InternationalrecommendationsonpediatricFBhavebeenpublishedby theEuropeanRespiratorySociety(ERS)andtheAmericanThoracicSocietyanddescribethe indications,thefacilities,andequipmentneededfortheprocedure,careoftheinstrumentsinvolved, techniques,andsuggestionsforsedationandpatientmanagement.(5-7) FBcanbeperformedfordiagnosticand/ortherapeuticpurposes.Itenablesanassessmentofthe airway'sanatomicalfeaturesandthecollectionofsamplesfromthedistalairways(bronchoalveolar lavage[BAL],bronchialbrushing,bronchialbiopsy)forpathologicalandmicrobiological examination.IndicationsfordiagnosticFB includestridor,persistent/re-currentwheezing,chronic cough(productiveorotherwise),recurrentpneumonia,suspectedforeignbodyaspiration, hemoptysisandpulmonaryhemorrhage,suspectedstructuralanomaliesorendobronchial lesions, radiographicabnormalities(atelectasis,recurrent/persistentconsolidations,atypicalandunknown infiltrates, localizedhyperinflation),monitoringoflungallograftorartificialairway,andobstructive sleepapnea)6,7). IndicationsfortherapeuticFB includerestoringairwaypatencyincasesofmucusplugsorblood clots,treatingalveolarfillingdisorders(alveolarproteinosisandlipidpneumonia),controlling hemorrhage,dilatingastenoticairway,andbronchoscopicintubation.(7) Theneedforgeneralanaesthesiainthesepatientsincreasestheproblemsofairwaybecauseof theneedtoshareanalreadycompromisedairwaywiththeendoscopist.Asimpleandsafemethod isdescribed.Generalanaesthesiaisinducedeitherbyintravenousorinhalationtechnique The childbreathesspontaneouslyviaamaskwithahighinspiredoxygenconcentrationandhalothane

a$thecordsaresprayedwithlignocaine.TheBodaisuction-safeswivel-Yconnector(Sontek MedicalInc.CatalogNo:SMI-1002)isaversatileplasticadapterwithstandard15mmfittingswhich sitswellbetweentheRendellBaker-SoucekmaskandtheAyre'sT-piece.(8,9) toevaluatetheindications&thefindingandtheadverseeventsofflexiblebronchoscopyat pediatric bronchoscopyunitatassuituniversitychildrenhospital

ELIGIBILITY:
Inclusion Criteria:

* Age group of children ≥1≤18 years

  * All children in pediatric bronchoscopy unit
  * Both sex
  * Children first guardians accepted to participate in the current study

Exclusion Criteria:

* age less than1year or more than 18 years

  * Children first guardians refused to participate in the current study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children in pediatric bronchoscopy unit
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
the adverse events of flexible bronchoscopy | baseline
  Severedesaturation(SaO2<80%)duringbronchoscopy